CLINICAL TRIAL: NCT00750438
Title: Increased Short Chain Fatty Acids in the Colon Are Associated With Improved Energy Homeostasis and Insulin Sensitivity.
Brief Title: Effect of Fibre Products on Appetite and Weight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 08/H0707/99
Record Dates: First submitted 2008-09-09; First posted 2008-09-10 (Estimated); Results first posted 2019-11-07 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Obesity
Keywords: Obesity; Short chain fatty acids; Appetite; Body weight; Insulin sensitivity; Propionate; Propionate ester
MeSH Terms: conditions — Obesity; Body Weight; Insulin Resistance | interventions — Inulin; Cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Propionate ester (Experimental)
  Interventions: Dietary Supplement: Propionate ester
- Fermentable control (Placebo Comparator)
  Interventions: Dietary Supplement: Inulin
- Non fermentable control (Placebo Comparator)
  Interventions: Dietary Supplement: Cellulose

INTERVENTIONS:
Dietary Supplement: Propionate ester — The subject will take propionate ester at the dose specified by the dose finding study, three times a day for 24 weeks
  Arms: Propionate ester
Dietary Supplement: Inulin — The subjects in this group will take inulin at a comparable dose, three times a day for 24 weeks
  Arms: Fermentable control
Dietary Supplement: Cellulose — The subjects in this group will take the non fermentable carbohydrate, cellulose, at a comparable dose for 24 weeks.
  Arms: Non fermentable control

SUMMARY:
This study explores the nutritional effects of fibre. Short chain fatty acid(SCFA), such as propionate, are produced through the fermentation of fibre in the bowel. SCFA are thought to have direct beneficial effects on the gut, appetite, weight and fat distribution. This study will look into these effects by conducting a dose finding study and then a randomised controlled study using healthy human volunteers.

DETAILED DESCRIPTION:
This is a dose finding study in healthy overweight to obese human volunteers (BMI 25- 35) to find the level of oral supplementation with propionate that increases plasma propionate levels to 10x the current normal plasma level and use this dose of propionate in a randomised, placebo controlled double bind study. This study will compare propionate with fermentable and non fermentable carbohydrate. The outcome measures for this study will include assessments of appetite with feeding studies, measurement of insulin sensitivity using hyperinsulinaemic euglycaemic clamps and assessment of adipose tissue distribution using MRI scans and adipose tissue biopsy to determine changes in proliferation and differentiation of adipocytes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers aged between 21 and 65 years

Exclusion Criteria:

* Weight change of more than 3kg in the preceding 2 months
* Current smokers
* Substance abuse
* Excess alcohol intake
* Pregnancy
* Diabetes
* Cardiovascular disease
* Cancer
* Gastrointestinal disease e.g. inflammatory bowel disease or irritable bowel syndrome
* Kidney disease
* Liver disease
* Pancreatitis
* Use of medications including: anti inflammatory drugs or steroids, cholesterol lowering medication, androgens, phenytoin, erythromycin or thyroid hormones.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-09 (Actual); Primary Completion 2012-07 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Frost, PhD, Principal Investigator — Imperial College London
Locations (1):
- Hammersmith Hospital, London, UK, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chambers ES, Viardot A, Psichas A, Morrison DJ, Murphy KG, Zac-Varghese SE, MacDougall K, Preston T, Tedford C, Finlayson GS, Blundell JE, Bell JD, Thomas EL, Mt-Isa S, Ashby D, Gibson GR, Kolida S, Dhillo WS, Bloom SR, Morley W, Clegg S, Frost G. Effects of targeted delivery of propionate to the human colon on appetite regulation, body weight maintenance and adiposity in overweight adults. Gut. 2015 Nov;64(11):1744-54. doi: 10.1136/gutjnl-2014-307913. Epub 2014 Dec 10. PMID 25500202
- [Derived] Byrne CS, Chambers ES, Alhabeeb H, Chhina N, Morrison DJ, Preston T, Tedford C, Fitzpatrick J, Irani C, Busza A, Garcia-Perez I, Fountana S, Holmes E, Goldstone AP, Frost GS. Increased colonic propionate reduces anticipatory reward responses in the human striatum to high-energy foods. Am J Clin Nutr. 2016 Jul;104(1):5-14. doi: 10.3945/ajcn.115.126706. Epub 2016 May 11. PMID 27169834

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Non fermentable arm not conducted
Groups:
- Inulin-control: Participants received inulin
- Inulin-propionate Ester: Participants received inulin-propionate ester
Period: Overall Study
Arm/Group | Inulin-control | Inulin-propionate Ester
Started | 31 | 29
Completed | 24 | 25
Not Completed | 7 | 4
Not completed — Protocol Violation | 4 | 1
Not completed — Physician Decision | 2 | 2
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inulin-control | Inulin-propionate Ester | Total
Number analyzed (Participants) | 24 | 25 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 25 | 49
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (1.5) | 55.3 (1.4) | 54 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 9 | 10 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 5 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 18 | 16 | 34
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 24 | 25 | 49
HbA1c [Mean (Standard Deviation); unit: mmol/mol] | 37.8 (0.5) | 38.2 (0.7) | 38 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Appetite_Food Intake
Description: The change in food intake following 24 weeks of supplementation
Time Frame: Baseline, 24 weeks
Measure: Mean (95% Confidence Interval); unit: kcal
Arm/Group | Inulin-control | Inulin-propionate Ester
Number analyzed (Participants) | 24 | 25
kcal
  Baseline | 678 [535 to 820] | 836 [724 to 948]
  24 weeks | 645 [514 to 776] | 763 [654 to 872]
Statistical Analysis 1: Comparison: Inulin-control vs Inulin-propionate Ester; Test type: Superiority; p = 0.972, Regression, Linear

2. Primary Outcome: Body Weight
Description: Body weight was measured in all subjects to the nearest 0.1 kg (Tanita BC-418MA) while subjects were wearing light clothing.
Time Frame: Baseline, 24 weeks
Measure: Mean (Standard Error); unit: kg
Arm/Group | Inulin-control | Inulin-propionate Ester
Number analyzed (Participants) | 24 | 25
kg
  Baseline | 91 (2.8) | 88.5 (2.9)
  24 weeks | 91.4 (3) | 87.5 (3)
Statistical Analysis 1: Comparison: Inulin-control; Baseline and 24 weeks; Test type: Superiority; p = 0.559, t-test, 2 sided
Statistical Analysis 2: Comparison: Inulin-propionate Ester; Baseline to 24 weeks; Test type: Superiority; p = 0.062, t-test, 2 sided
Statistical Analysis 3: Comparison: Inulin-control vs Inulin-propionate Ester; Test type: Superiority; p = 0.099, Regression, Linear

3. Primary Outcome: Body Weight - Number of Participants Gained ≥3% of Their Baseline Body Weight
Description: as for outcome 2
Time Frame: Baseline, 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Inulin-control | Inulin-propionate Ester
Number analyzed (Participants) | 24 | 25
Participants | 6 | 1
Statistical Analysis 1: Comparison: Inulin-control vs Inulin-propionate Ester; Test type: Superiority; p = 0.036, Regression, Linear

4. Secondary Outcome: Adipose Tissue Distribution - Intra-abdominal Adipose Tissue
Description: Body composition was assessed using MRI and MR spectroscopy (MRS), expressed as a percentage of total adipose tissue content.
Time Frame: 24 weeks
Population: MRS data could not be collected in 17 subjects, due to metal implants (n=8) and claustrophobia (n=9).
Measure: Mean (Standard Error); unit: percentage of total adipose tissue
Arm/Group | Inulin-control | Inulin-propionate Ester
Number analyzed (Participants) | 15 | 17
percentage of total adipose tissue
  Baseline | 10.6 (1.3) | 13.2 (1.2)
  24 weeks | 11.1 (1.4) | 13.1 (1.1)
Statistical Analysis 1: Comparison: Inulin-control; Baseline to 24 weeks; Test type: Superiority; p = 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Inulin-propionate Ester; Baseline to 24 weeks; Test type: Superiority; p = 0.723, t-test, 2 sided
Statistical Analysis 3: Comparison: Inulin-control vs Inulin-propionate Ester; Test type: Superiority; p = 0.027, Regression, Linear

5. Secondary Outcome: Insulin Sensitivity - HOMA IR
Description: The homeostatic model assessment (HOMA) is a method used to quantify insulin resistance and beta-cell function.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: percentage of Beta Cell Function
Arm/Group | Inulin-control | Inulin-propionate Ester
Number analyzed (Participants) | 24 | 25
percentage of Beta Cell Function
  Baseline | 2.7 (0.3) | 2 (0.2)
  24 weeks | 2.3 (0.2) | 2 (0.2)
Statistical Analysis 1: Comparison: Inulin-control; Test type: Superiority; p = 0.372, t-test, 2 sided
Statistical Analysis 2: Comparison: Inulin-propionate Ester; Test type: Superiority; p = 0.644, t-test, 2 sided
Statistical Analysis 3: Comparison: Inulin-control vs Inulin-propionate Ester; Test type: Superiority; p = 0.549, Regression, Linear

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Inulin-control | Inulin-propionate Ester
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/29
Other Adverse Events (participants affected / at risk) | 14/31 | 5/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inulin-control (N=31) | Inulin-propionate Ester (N=29)
Stomach discomfort (Gastrointestinal disorders) | 8 (8) | 1 (1)
Bloating (Gastrointestinal disorders) | 8 (8) | 3 (3)
Flatulence (Gastrointestinal disorders) | 14 (14) | 5 (5)
Heartburns (Gastrointestinal disorders) | 3 (3) | 2 (2)
Belching (Gastrointestinal disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes